CLINICAL TRIAL: NCT05812703
Title: What Objective Changes Occur With Behavioral Treatment: Evaluating Biometrics and Self -Reported Health Measures of Adult Patients Receiving Behavioral Treatments With Chronic Pain
Brief Title: Biometrics and Self-reported Health Changes in Adults Receiving Behavioral Treatments for Chronic Pain
Status: Not yet recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Heather Poupore-King, Clinical Associate Professor, Stanford University
Other Study IDs: 66952
Record Dates: First submitted 2023-03-31; First posted 2023-04-14 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Chronic Pain; Sedentary Time
Keywords: movement; behavioral treatments; biometrics; chronic pain
MeSH Terms: conditions — Chronic Pain; Sedentary Behavior | interventions — Cognitive Behavioral Therapy; Acceptance and Commitment Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Biospecimen Retention: Samples Without DNA — HR variability, Activity (steps), Sedentary time, Sleep Stages (REM, light, deep)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Behavioral Group Treatment (Cognitive Behavioral Therapy CBT + Movement): Cognitive Behavioral Therapy Group led by a psychologist to learn pain coping skills, with gentle movement component of duration from 45 minutes to 60 minutes under a licensed Healthcare provider (PT or OT).
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Behavioral Group Treatment (ACT) only: Acceptance and Commitment Therapy Group led by a psychologist to learn skills to change their relationship with pain to decrease pain's impact on their life.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)
- Behavioral Group Treatment (ACT + Movement)- Back in ACTion: Acceptance and Commitment Therapy Group led by a psychologist to learn skills to change their relationship with pain to decrease pain's impact on their life and improve willingness to engage in valued activities. Movement component to last from with intense and gentle movement sessions with a total movement time of 90 minutes - 2 hours led by licensed health care provider a PT or OT.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT); Behavioral: Moderate to high Intensity Group Exercise

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — The participants will attend one of the behavioral group treatments programs offered by the Stanford Pain Management Center. This class may be held online via Zoom, or in person based at the Stanford Pain Management Center. The class may be recorded for training purposes. No names or images/faces will be recorded for privacy reasons. The behavioral groups are 3 types, with or without exercise/movement. Current Evidence Based treatments that are provided as standard practice include: Cognitive Behavioral Therapy Group, with movement, Acceptance and Commitment Therapy Group, with or without movement. Group participants will learn different skills in each group and develop a personalized plan to use the skills after group ends. At the end of group participants will be given an anonymous survey about the class to evaluate satisfaction of the treatment. Movement in this portion of class is designed to low impact and restorative/gentle, with no significant increases in HR > 50% HRmax.
  Other Names: Pain Coping Skills; Group Movement
  Groups: Behavioral Group Treatment (Cognitive Behavioral Therapy CBT + Movement)
Behavioral: Acceptance and Commitment Therapy (ACT) — ACT is a 6 week behavioral group program led by a psychologist to improve psychological flexibility and reduce pain interference in patients with chronic pain.
  Groups: Behavioral Group Treatment (ACT + Movement)- Back in ACTion; Behavioral Group Treatment (ACT) only
Behavioral: Moderate to high Intensity Group Exercise — Group exercise led by supervised clinician with Cardiovascular focus to increase HR into zones to see adaptations to improve cardiovascular fitness.
  Groups: Behavioral Group Treatment (ACT + Movement)- Back in ACTion

SUMMARY:
The study will provide important information regarding the biometric changes that occur in behavioral treatments for chronic pain and explore the additional impact of integrated movement and supervised exercise. The goal of this clinical trial is to determine if pain rehabilitation programs have impacts on physical function in patient reported outcomes and objective measures of physical activity or sedentary time with a wearable Fitbit. Additionally, we will examine the associations between movement, pain acceptance, and related health factors, such as pain severity, sleep, functional status, depression, and anxiety. The addition of biometric data will allow for further investigation of the association between objective measures and patient self-report measures.

DETAILED DESCRIPTION:
Chronic pain has high impact on societal function as well as an individual person's mood, physical function, disability, and quality of life and their health. The purpose of the study is to collect objective outcome measures on movement, activity, biometrics and patient reported outcome measures for participants of behavioral treatment groups of 6-8 weeks duration at Stanford Pain Management Center. Group participants learn skills and develop a personalized plan to use the skills throughout the program. The study will follow participants with a removable wearable device on the wrist for 2 weeks pre group to establish movement activity baselines, during the group intervention (6-8 weeks) and 2 weeks post group to determine which groups have benefits across various aspects of health including: sleep, psychological processes of pain acceptance, physical mobility, quality of life and the impact of supervised movement and physical activity in the treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18+
2. Non-cancer chronic pain (pain that occurs on at least half of the days of 6 months or more)
3. English fluency
4. Ability to attend >70% treatment sessions to ensure active treatment is delivered

Exclusion Criteria:

1. Cognitive impairment, non-English speaking, or psychological factors that would preclude comprehension of material and/or full participation in the study.
2. Participants with acute cauda equina syndrome
3. Inability to complete a 6 minute walk test without LOB

3) Chronic pain as explained by inflammatory disease

For the movement-based portions of group:

Exclusion: For our CBT + Movement (low intensity/ restorative) movement group: Patient must be able to sit upright for 20 minutes without loss of balance or upper extremity (UE) assistance. Inability to sit without use of UE support would be excluded. This ensures safety that the participant can completed the adapted movement program without risk of falls. HR will not be elevated > 50% HRmax in these restorative movement classes.

Exclusion criteria for the Back in ACTion (higher intensity) movement group is inability to complete a 6-minute walk test safely or without loss of balance, as this poses a fall risk that requires individual assistance throughout the class, or medical exclusion from cardiovascular exercise over 50% HRmax, as HR will be elevated to 50-70% HR max in these classes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — We will include self-reported gender preferences
Study Population: Participants with chronic pain
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-09-27 (Estimated); Primary Completion 2025-10-25 (Estimated); Study Completion 2026-04-25 (Estimated)

PRIMARY OUTCOMES:
Change in sedentary behavior time | Pre intervention (baseline), and post intervention (at 10 weeks)
  Sedentary behavior is defined as any waking behavior such as sitting or leaning with an energy expenditure of 1.5 metabolic equivalent task (MET) or less

SECONDARY OUTCOMES:
HF-Heart rate variability | Pre intervention (baseline), end of treatment session (week 6), and post intervention (at 10 weeks)
  Heart rate variability (per participant) is where the amount of time between your heartbeats fluctuates slightly. Even though these fluctuations are undetectable except with specialized devices, they can still indicate current or future health problems, including heart conditions and mental health issues like anxiety and depression. Heart rate variability (in milliseconds) has no standard reference range. HF is the high frequency band of HRV.
Sleep Duration | Pre intervention (baseline), end of treatment session (week 6), and post intervention (at 10 weeks)
  Amount of time asleep per "night cycle"
Daily Step Count | Pre intervention (baseline), end of treatment session (week 6), and post intervention (at 10 weeks)
  Amount of steps occurring in a 24 hour day
Pain Catastrophizing | Pre intervention (baseline), and post intervention (at 10 weeks) and 6 months follow up (post group)
  13-item self-report measure designed to assess catastrophic thinking related to pain among adults. The score ranges from 0-52, where higher scores indicate greater pain catastrophizing.
PROMIS Depression Score | Pre intervention (baseline), and post intervention (at 10 weeks),and 6 months follow up (post group)
  Self reported Questionnaires to assess depression. Patient-Reported Outcomes Measurement Information System (PROMIS) - Depression use a T-score metric, and the scores range from 10T to 85T, with the population mean score of 50T (SD of 10). Higher T scores would indicate worse symptom in each domain.
PROMIS Anxiety Score | Pre intervention (baseline), and post intervention (at 10 weeks),and 6 months follow up (post group)
  Self reported Questionnaires to assess anxiety. Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety measures use a T-score metric, and the scores range from 10T to 85T, with the population mean score of 50T (SD of 10). Higher T scores would indicate worse symptom in each domain.
PROMIS Sleep Disturbance Score | Pre intervention (baseline), and post intervention (at 10 weeks),and 6 months follow up (post group)
  Self reported Questionnaires to assess sleep quality. Patient-Reported Outcomes Measurement Information System (PROMIS) , Sleep Disturbance use a T-score metric, and the scores range from 10T to 85T, with the population mean score of 50T (SD of 10). Higher T scores would indicate worse symptom in each domain.
PROMIS Physical Function Score | Pre intervention (baseline), and post intervention (at 10 weeks),and 6 months follow up (post group)
  Self reported Questionnaires to assess physical function/mobility. Patient-Reported Outcomes Measurement Information System (PROMIS) physical function measures use a T-score metric, and the scores range from 10T to 85T, with the population mean score of 50T (SD of 10). Higher T scores would indicate worse symptom in each domain.
PROMIS Pain Interference Score | Pre intervention (baseline), and post intervention (at 10 weeks),and 6 months follow up (post group)
  Self-reported Questionnaires to assess pain interference. Patient-Reported Outcomes Measurement Information System (PROMIS), pain interference, and physical function measures use a T-score metric, and the scores range from 10T to 85T, with the population mean score of 50T (SD of 10). Higher T scores would indicate worse symptom in each domain.
Duration of Heart Rate in Exercise Zones (50-70% HRMax) (during exercise) | Pre intervention (baseline), and post intervention (at 10 weeks)
  The time in a 24 hour period that the participant has an elevated heartrate for sustained duration indicating exercise.
  We would want to increase our amount of time (minutes) in HRzones to indicate more time spend in active exercise during the movement portions of the interventions.
Average Resting Heartrate | Pre intervention (baseline), end of treatment session (week 6), and post intervention (at 10 weeks)
  A 2013 study in the journal Heart tracked the cardiovascular health of about 3,000 men for 16 years and found that a high resting heart rate was linked with lower physical fitness and higher blood pressure, body weight, and levels of circulating blood fats. The researchers also discovered that the higher a person's resting heart rate, the greater the risk of premature death. Specifically, an RHR between 81 and 90 doubled the chance of death, while an RHR higher than 90 tripled it.
  A low resting heart rate often suggests greater physical fitness. A reduction in average resting heart rate would indicate improvement in CV fitness for our treatment interventions.
Physical Activity Vital Sign | Pre intervention (baseline), end of treatment session (week 6), and post intervention (at 10 weeks)
  the subjective measure of minutes a person is physically active in a week (in minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Heather King, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Pain Management Clinic, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] You DS, Ziadni MS, Cooley CE, Talavera DC, Mackey SC, Poupore-King H. Effectiveness of a multidisciplinary rehabilitation program in real-world patients with chronic back pain: A pilot cohort data analysis. J Back Musculoskelet Rehabil. 2021;34(6):965-973. doi: 10.3233/BMR-200305. PMID 34151829
- [Background] Neumann A, Hampel P. Long-term effects of rehabilitation and prevention of further chronification of pain among patients with non-specific low back pain. J Back Musculoskelet Rehabil. 2022;35(6):1257-1268. doi: 10.3233/BMR-210221. PMID 35754259
- [Background] Pears S, Sutton S. Effectiveness of Acceptance and Commitment Therapy (ACT) interventions for promoting physical activity: a systematic review and meta-analysis. Health Psychol Rev. 2021 Mar;15(1):159-184. doi: 10.1080/17437199.2020.1727759. Epub 2020 Feb 17. PMID 32036768
- [Background] Mercer K, Li M, Giangregorio L, Burns C, Grindrod K. Behavior Change Techniques Present in Wearable Activity Trackers: A Critical Analysis. JMIR Mhealth Uhealth. 2016 Apr 27;4(2):e40. doi: 10.2196/mhealth.4461. PMID 27122452
- [Background] Shaffer F, Ginsberg JP. An Overview of Heart Rate Variability Metrics and Norms. Front Public Health. 2017 Sep 28;5:258. doi: 10.3389/fpubh.2017.00258. eCollection 2017. PMID 29034226
- [Background] Karayannis NV, Sturgeon JA, Kemani MK, Mackey SC, Greco CM, Wicksell RK, McCracken LM. Pain acceptance and psychological inflexibility predict pain interference outcomes for persons with chronic pain receiving pain psychology. Scand J Pain. 2023 Feb 7;23(3):464-475. doi: 10.1515/sjpain-2022-0107. Print 2023 Jul 26. PMID 36745187